CLINICAL TRIAL: NCT04161794
Title: Multimodal Intervention (Dietary Counselling, Fish Oil and Physical Training) for Patients With Non-small Cell Lung Cancer, a Feasibility Study
Brief Title: Multimodal Intervention for Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Randi Tobberup, Ph.D. student, Aalborg University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LUCANU-2
Record Dates: First submitted 2019-09-24; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Cachexia; Cancer
Keywords: cachexia; cancer; multimodal intervention
MeSH Terms: conditions — Cachexia; Neoplasms | interventions — Combined Modality Therapy

STUDY DESIGN:
Intervention Model Description: This is a single arm intervention study, comparing the results to that of a historical control Group.
Masking Description: Non-randomised
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 2 g EPA/DHA via fish oil daily Regular dietary counselling Twice weekly strength and cardiovascular exercise
  Interventions: Other: multimodal
- Historical control group (No Intervention): Standard of Care

INTERVENTIONS:
Other: multimodal — 2 g EPA/DHA as fish oil, repeated dietary counselling and twice weekly 2 x exercises
  Arms: Intervention group

SUMMARY:
A single-arm intervention study assessing the feasibility of a multimodal intervention of management of cancer cachexia in patients with non-small cell lung cancer during primary anti-neoplastic treatment. The effects of the intervention is compared to a historical control group

DETAILED DESCRIPTION:
In a single arm intervention study, we will provide a multimodal intervention consisting of dietary counselling, physical exercises plan as well as fish oil.

The target of the dietary counselling is:

* 30 kcal/kg/d (in patients with BMI <30) or 25 kcal/kg/d (in patients with BMI => 30)
* at least 1.0 g protein/kg/d
* three daily meals of at least 20 g of protein
* restrict overnight fasting to a maximum of 11 hours

The initial dietary counselling is at the first cycle of anti-neoplastic treatment. The patient will be provided an individual plan to meet the dietary targets tailored to the individual preferences and symptoms. At every cycle of anti-neoplastic treatment, the plan will be adjusted if needed. At every week the patients will be prompted by telephone to comply with the dietary plan.

The physical exercise consists of two exercises:

* strength training: a progressive sit-to-stand exercise which is a lower extremity exercise.
* cardio-vascular training: a progressive brisk walking plan. Patients are prompted to execute both exercises twice weekly. The individual targets are set at the first cycle of anti-neoplastic treatment and adjusted during the trial.

Fish oil:

The patients are instructed to ingest 10g of liquid fish oil (consisting of 2 g EPA/DHA) or 8 capsules of fish oil (consisting of 2 g EPA/DHA)

ELIGIBILITY:
Inclusion Criteria:

* histopathologically or cytologically verified with NSCLC
* inoperable tumour, candidates for, but naïve to or no systemic anti-neoplastic treatment the previous two years
* commence first line of chemotherapy (carboplatin/vinorelbin, cisplatin/vinorelbin) with or without radiation therapy or pembrolizumab
* performance status ≤2 (Eastern Cooperative Oncology Group)
* age >18 and provided oral
* written consent

Exclusion Criteria:

* excessive alcohol or drug abuse
* incapable to follow the intervention (i.e. cognitive problems or unable to walk) were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility, recruitment rate | 9 months
  Recruitment rate is measured by dividing the number of patients consented by the number of patients screened
Feasibility, retention rate | 9 months
  Retention rate is measured by dividing the number of patients completing the trial with the number of patients consented
Feasibility, compliance | 9-18 weeks
  The overall compliance was defined successful if at least half of the included patients reached at least 75 % of the nutrient target, consumed at least 75 % of the fish oil and conducted at least 50 % of the physical exercises

SECONDARY OUTCOMES:
Predictive and prognostic factors of change in skeletal muscle | 9-18 weeks
  Change in skeletal muscle was measured using CT scans, analysed at the 3rd lumbar vertebra, expressed as actual change in square centimeter. Using an ordinal logistic regression model, patients were ordered in three Groups (muscle wasting: loss of at least 6 cm^2 ; muscle maintenance: +/- 5.9 cm^2; muscle gain: gain of at least 6.0 cm^2). The baseline variables included in the model are age, gender, tumor stage, type of treatment, performance status, inflammatory score (mGPS) and cachexia. The possible prognostic factors included in the model is change in body weight, adherence to the anti-neoplastic treatment plan, treatment response, compliance to the multimodal intervention, number of Nutrition impact symptoms, days in between CT scans, energy and protein intake.
Group difference in body weight | 9-18 weeks
  The change in body weight (measured at baseline and at the end of the trial using body weight scales, expressed as %
Group difference in skeletal muscle | 9-18 weeks
  Change in skeletal muscle (measured using CT scans, expressed as actual muscle change at the 3rd lumbar vertebra in mean (SD) cm^2
Proportion of patients gaining, maintaining and wasting of skeletal muscle | 9-18 weeks
  expressed as number of patients. Gaining defined as at least +6 Square centimeter skeletal muscle. Maintaining defined as: +/- 5.9 Square centimeter skeletal muscle. Wasting defined as: at least -6 Square centimeter skeletal muscle
Change in physical function | 9-18 weeks
  assessed by timed-up-and-go test (expressed in number of seconds) and assessed by 30 seconds sit-to-stand test (expressed as number of stands).

CONTACTS AND LOCATIONS:
Overall Officials: Mette Holst, PhD, Study Chair — Aalborg University Hospital
Locations (1):
- Aalborg Univeristy Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tobberup R, Carus A, Rasmussen HH, Falkmer UG, Jorgensen MG, Schmidt EB, Jensen NA, Mark EB, Delekta AM, Antoniussen CS, Bogsted M, Holst M. Feasibility of a multimodal intervention on malnutrition in patients with lung cancer during primary anti-neoplastic treatment. Clin Nutr. 2021 Feb;40(2):525-533. doi: 10.1016/j.clnu.2020.05.050. Epub 2020 Jun 9. PMID 32600857